CLINICAL TRIAL: NCT00996229
Title: Phase IV Interventional Study: Effects of Dietary Interventions on Brain Functions in Healthy Elderly People
Brief Title: Effects of Dietary Interventions on the Aging Brain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Floel, Prof. Dr. med. Agnes Flöel, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ernaehrung-Neuromod 02
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Diet; elderly; cognition; prevention; cognitive decline; Lifestyle
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Caloric Restriction; Docosahexaenoic Acids; Fish Oils; Resveratrol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Caloric restriction + placebo supplementation (Experimental)
  Interventions: Behavioral: Caloric restriction; Dietary Supplement: Placebo
- Omega-3 supplementation (Experimental)
  Interventions: Dietary Supplement: Omega-3 (fish oil capsules)
- Placebo supplementation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Resveratrol supplementation (Experimental)
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Behavioral: Caloric restriction — 20-30% CR for 6 months
  Arms: Caloric restriction + placebo supplementation
Dietary Supplement: Omega-3 (fish oil capsules) — 2g/day DHA/EPA capsules for 6 months
  Arms: Omega-3 supplementation
Dietary Supplement: Placebo — Daily corn oil capsules for 6 months
  Arms: Caloric restriction + placebo supplementation; Placebo supplementation
Dietary Supplement: Resveratrol — daily resveratrol for 6 months
  Arms: Resveratrol supplementation

SUMMARY:
The researchers will investigate whether caloric restriction or dietary supplementation could provide positive effects on general brain functions in healthy elderly people.

DETAILED DESCRIPTION:
The age-related degradation of cognitive functions even to the point of neurodegenerative disorders such as Alzheimer's disease are a growing public-health concern with devastating effects.

Referring to animal data, empirical studies, and pilot human trials, a healthy diet rich in unsaturated fatty acids and low in calories should improve cognitive functions such as learning and memory. To test this hypothesis, the researchers study general brain functions in healthy elderly subjects (50-80 years old) during a short term diet.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* 50-80 years old
* moderate to heavy weight (BMI 25-30)
* must be able to change diet/take supplements at home

Exclusion Criteria:

* diabetes
* younger than 50 years
* BMI < 25
* psychiatric medication
* severe disease
* MMSE < 26
* eating disorders

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Auditory verbal Learning Task | Baseline (timepoint 0), after 6 months (timepoint 6 months)

SECONDARY OUTCOMES:
Functional/Structural brain changes | Baseline (timepoint 0), after 6 months (timepoint 6 months)
Plasma biomarkers | Baseline (timepoint 0), after 6 months (timepoint 6 months)f intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Professor, Study Chair — Charite University, Berlin, Germany; Veronica Witte, Dr, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Neurology, Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany